CLINICAL TRIAL: NCT01520571
Title: Do We Need Computer Assistance To Improve the Survival of Primary Total Knee Arthroplasty. A Minimum Ten Years Follow-up
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, Young Hoo Kim, Professor and Director, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Computer Assistance TKA
Record Dates: First submitted 2012-01-19; First posted 2012-01-30 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Osteoarthritis
Keywords: Computer Assistance; Total Knee Arthroplasty; conventional
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Computer Assistance TKA (Active Comparator): Non-Computer Assistance TKA
  Interventions: Procedure: Non-Computer Assistance TKA
- Computer Assistance TKA (Experimental): Computer Assistance TKA
  Interventions: Procedure: Computer Assistance TKA

INTERVENTIONS:
Procedure: Non-Computer Assistance TKA — Non-Computer Assistance Total Knee Arthroplasty
  Other Names: Non-Computer Assistance Total Knee Arthroplasty
  Arms: Non-Computer Assistance TKA
Procedure: Computer Assistance TKA — Computer Assistance Total Knee Arthroplasty
  Other Names: Computer Assistance Total Knee Arthroplasty
  Arms: Computer Assistance TKA

SUMMARY:
The investigators asked: (1) Do computer-assisted total knee arthroplasty (TKAs) provide better alignment and clinical function? (2) Do computer-assisted TKAs provide better survivorship of implants and less complication? and (3) Do correction of the mechanical axis of the lower limb to within 3° of neutral is a prognostic marker for late revision surgery due to aseptic loosening?

DETAILED DESCRIPTION:
Computer-assisted total knee arthroplasty (TKA) is reported to improve the overall accuracy of positioning of the femoral and tibia components. However, an acceptable target for alignment remains a matter for debate. A mechanical axis within 3° of neutral axis has been used as the primary outcome measure in many clinical trials comparing computer-assisted- and conventional TKA. However, the evidence supporting this arbitrary value is unreliable because previous reports are limited by their small sample size, inadequate radiographs, short follow-up and lack of clarity when defining a margin of accuracy.

ELIGIBILITY:
Inclusion Criteria:

* End stage osteoarthritis of the knee joint who require total knee arthroplasty with bilateral lesions.

Exclusion Criteria:

* Inflammatory disease
* patient with other Lower extremity disease which may affect functional outcome
* Neurologic disease effecting patients lower extremity
* Revision surgery
* Patient not medically cleared for bilateral surgery

Ages: 49 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2000-01; Primary Completion 2001-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Improvement in Knee Society Knee Score | 10.5 years
  change in knee score will be compared with initial score, until follow up of 10.5 years

SECONDARY OUTCOMES:
Improvement in the range of motion | 10.5 years
  change in the range of motion of knee joint will be compared with the initial value, until follow up of 10.5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoo Kim, MD, Study Director — Ewha Womans University School of Medicine
Locations (1):
- Ewha Womans University Mokdong Hosptial, Seoul, South Korea